CLINICAL TRIAL: NCT06615700
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of NA-931 in Overweight/Obese Participants and in Patients With Type 2 Diabetes Mellitus
Brief Title: Phase 1 to Study Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NA-931 in Obese Participants and Patients With Type 2 Diabetes Mellitus
Acronym: T2DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomed Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA-931-50
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Overweight or Obesity; Type 2 Diabetes
Keywords: NA-931, obesity, Type 2 Diabetes, Biomed Industries, Inc
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant Group/Arm- NA-931 (Experimental): Experimental: NA-931 Capsule of NA-931 intervention
  Interventions: Drug: NA-931
- Participant Group/Arm- Placebo (Placebo Comparator): Placebo Comparator: Placebo Capsule of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NA-931 — NA-931 is a quadruple receptor agonist for weight loss
  Other Names: NA-931 is a quadruple receptor agonist
  Arms: Participant Group/Arm- NA-931
Drug: Placebo — Placebo of NA-931
  Other Names: Placebo of NA-931
  Arms: Participant Group/Arm- Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, dose escalation, first in human study designed to assess the safety and tolerability, pharmacokinetics, and pharmacodynamics of NA-931 when administered as single and multiple-ascending doses in overweight/obese participants and as multiple doses in patients with T2DM.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, dose escalation, first in human study designed to assess the safety and tolerability, pharmacokinetics, and pharmacodynamics of NA-931 when administered as single and multiple-ascending doses in overweight/obese participants and as multiple doses in patients with Type 2 Diabetes Mellitus.

NA-931 is a Quadruple Receptor Agonist for Insulin Like Growth Factor 1 (IGF-1), Glucagon-like Peptide-1 (GLP-1), Gastric Inhibitory Polypeptide (GIP) and Glucagon.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18-65 years old, inclusive
* BMI of 25 - 40, inclusive
* Stable body weight for two months
* Participants must be capable of giving signed informed consent
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other clinical study procedures
* Willing to comply with contraception requirements

Exclusion Criteria:

* History of significant medical conditions and malignancy
* Uncontrollable hypertension
* History of alcoholism or drug addiction within 1 year prior to Screening
* Current or recent participation in an investigational clinical trial
* Any surgical or medical condition (active or chronic) that may interfere with IP distribution, metabolism, excretion, or drug absorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events in NA-931 participants | 28 days
  To evaluate the safety and tolerability of NA-931

SECONDARY OUTCOMES:
Maximum observe drug concentration (Cmax) of NA-931 | 28 days
  Pharmacokinetics (PK) Cmax
Effect of a High-Fat Meal on Plasma Concentration of NA-931 | 28 days
  Determine the effect of a high-fat meal on the Pharmacokinetics of NA-931following a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Tran, PhD, Study Director — Biomed Industries, Inc.
Locations (2):
- Australia (2):
  - Biomed Industries Pty Limited- Clinical Testing Site 1, Camperdown, New South Wales
  - Biomed Industries, Pty Limited Testing Site 2, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No